CLINICAL TRIAL: NCT06437236
Title: Comparative Study Between Intravenous Granisetron and Ondansetron on Their Effect on Hemodynamics and Shivering After Spinal Anesthesia in Elective Cesarean Delivery : A Randomized Double-Blind Study
Brief Title: Comparative Study Between Intravenous Granisetron and Ondansetron on Their Effect on Hemodynamics and Shivering After Spinal Anesthesia in Elective Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrady Abdelaziz, resident at Anesthesiology, Surgical Intensive Care and Pain Medicine department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-24-04-012MS
Record Dates: First submitted 2024-05-20; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hemodynamic Instability and Shivering
MeSH Terms: interventions — Ondansetron; Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): will receive ondansetron 4mg diluted in normal saline,The total volume of the solution infused will kept at 10 mL.
  After preloading, patients in the respective group will receive the infusion of the study drug over 1 minute just 5 minutes before performing the subarachnoid block.
  Interventions: Drug: ondansetron
- group B (Active Comparator): will receive granisetron 1mg diluted in normal saline.The total volume of the solution infused will kept at 10 mL.
  After preloading, patients in the respective group will receive the infusion of the study drug over 1 minute just 5 minutes before performing the subarachnoid block.
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: ondansetron — Group A will receive ondansetron 4mg diluted in normal saline,The total volume of the solution infused will kept at 10 mL.
  After preloading, patients in the respective group will receive the infusion of the study drug over 1 minute just 5 minutes before performing the subarachnoid block
  Arms: Group A
Drug: granisetron — Group B will receive granisetron 1mg diluted in normal saline.The total volume of the solution infused will kept at 10 mL.
  After preloading, patients in the respective group will receive the infusion of the study drug over 1 minute just 5 minutes before performing the subarachnoid block
  Arms: group B

SUMMARY:
Spinal anesthesia is commonly used in cesarean section surgeries . The most important adverse effects of spinal anesthesia are hypotension and bradycardia caused by sympathetic blockade, with an incidence of about 55-100% . However, blocking the venous return by the gravid uterus increases the risk of hypotension. Spinal anesthesia-induced hypotension is commonly associated with uncomfortable symptoms, such as shivering , nausea and vomiting, in the mother. Prolonged maternal hypotension may lead to serious maternal adverse effects, such as cardiovascular collapse, loss of consciousness, apnea, and aspiration of gastric contents. In addition, uteroplacental blood flow decreases in cases of sustained hypotension and detrimental neonatal effects, such as fetal acidosis and fetal death, may occur. Preventing spinal anesthesia-induced hypotension during cesarean section is essential for the well-being of both the mother and neonate.

Also, Shivering often happens after spinal anesthesia. Shivering is an unconscious and rhythmic movement involving several groups of muscles. The increase of muscle activity generates the elevation of oxygen consumption, lactic acidosis, and carbon dioxide production In recent years, researchers have focused on the effects of the Bezold-Jarisch reflex (BJR) . This reflex includes a triad of bradycardia, hypotension, and apnea. Researchers have suggested that serotonin and 5-hydroxytryptamine 3 (5-HT3) receptors play an important role in the occurrence of the BJR after spinal anesthesia . The 5-HT3 receptors are present in the heart, lung, and spine. Diminished venous return caused by spinal anesthesia stimulates the cardiac chemoreceptors, and parasympathetic activity increases, which results in bradycardia and hypotension . Studies have suggested that the use of 5-HT3 antagonists may attenuate spinal anesthesia-induced hypotension, thus inhibiting peripheral vasodilatation, alleviating the BJR, and increasing venous return to the heart . Ondansetron is a commonly used 5-HT3 receptor antagonist, and its peak plasma concentration occurs within 30 min following IV injection. Granisetron is a new 5-HT3 receptor antagonist, and the onset of action occurs 30 min following its IV administration [

ELIGIBILITY:
Inclusion Criteria:

* All parturient who underwent elective caesarean delivery under spinal anesthesia will be included in this study

Exclusion Criteria:

* 1. Patient refusal 2. Patient with significant neurological , psychological disease 3. patient known allergy to ondansetron or granisetron, 4. patients receiving serotonin agonists or antagonists, 5. patient ischemic heart disease, chronic hypertension or pregnancy induced hypertension

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure mesurment in mmhg | 6 months
  a comparison of change in Blood pressure among groups

SECONDARY OUTCOMES:
incidece of shivering or not | 6 months
  will include detect difference among groups incidece of shivering or not

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JE, George RB, Habib AS. Spinal-induced hypotension: Incidence, mechanisms, prophylaxis, and management: Summarizing 20 years of research. Best Pract Res Clin Anaesthesiol. 2017 Mar;31(1):57-68. doi: 10.1016/j.bpa.2017.01.001. Epub 2017 Jan 8. PMID 28625306
- [Background] Kinsella SM, Tuckey JP. Perioperative bradycardia and asystole: relationship to vasovagal syncope and the Bezold-Jarisch reflex. Br J Anaesth. 2001 Jun;86(6):859-68. doi: 10.1093/bja/86.6.859. PMID 11573596
- [Background] Ortiz-Gomez JR, Palacio-Abizanda FJ, Morillas-Ramirez F, Fornet-Ruiz I, Lorenzo-Jimenez A, Bermejo-Albares ML. The effect of intravenous ondansetron on maternal haemodynamics during elective caesarean delivery under spinal anaesthesia: a double-blind, randomised, placebo-controlled trial. Int J Obstet Anesth. 2014 May;23(2):138-43. doi: 10.1016/j.ijoa.2014.01.005. Epub 2014 Feb 4. PMID 24631057
- [Background] Yeoh SB, Leong SB, Heng AS. Anaesthesia for lower-segment caesarean section: Changing perspectives. Indian J Anaesth. 2010 Sep;54(5):409-14. doi: 10.4103/0019-5049.71037. PMID 21189878